CLINICAL TRIAL: NCT06430671
Title: Multicenter, Phase Ib/IIa Study on the Safety and Efficacy of Autologous Peptide-coupled Red Blood Cells in Patients With Relapsing Remitting Multiple Sclerosis - RED4MS Trial
Brief Title: Peptide-coupled Red Blood Cells for the Treatment of Multiple Sclerosis
Acronym: RED4MS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cellerys AG (Industry)
Collaborators: Novartis (Industry); Scope International AG (Industry); Tetec AG (Industry); Jung Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MSB-IG-H-2101
Record Dates: First submitted 2024-05-06; First posted 2024-05-28 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Relapsing-remitting Multiple Sclerosis (RRMS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Intervention Model Description: Individual patients will be assigned to three dose groups. Patients will be allocated in the low, medium, high dose group according to the order of recruitment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CLS12311 low (Experimental): Low dose CLS12311
  Interventions: Drug: CLS12311 low; Drug: uncoupled RBCs
- CLS12311 medium (Experimental): Medium dose CLS12311
  Interventions: Drug: CLS12311 medium; Drug: uncoupled RBCs
- CLS12311 high (Experimental): High dose CLS12311
  Interventions: Drug: CLS12311 high

INTERVENTIONS:
Drug: CLS12311 low — Peptide-coupled Red Blood Cells (RBCs)
  Arms: CLS12311 low
Drug: CLS12311 medium — Peptide-coupled Red Blood Cells (RBCs)
  Arms: CLS12311 medium
Drug: CLS12311 high — Peptide-coupled Red Blood Cells (RBCs)
  Arms: CLS12311 high
Drug: uncoupled RBCs — autologous Red Blood Cells (RBCs)
  Arms: CLS12311 low; CLS12311 medium

SUMMARY:
RED4MS is a clinical trial to assess the safety and tolerability of autologous peptide coupled red blood cells (CLS12311) in patients with relapsing remitting multiple sclerosis (RRMS). CLS12311 consists of autologous red blood cells (RBCs) coupled with antigenic peptides and aims to treat RRMS by induction of antigen-specific immune tolerance.

DETAILED DESCRIPTION:
The RED4MS trial is designed as an open-label, dose-escalation phase Ib study, enrolling 9 RRMS patients in three ascending dose groups. The first patient (sentinel) in each dose group will receive one cycle of the therapy, while the remaining patients will receive two treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

1. RRMS according to the 2017 McDonald criteria
2. Male or female patients (assigned at birth) aged 18-55 years inclusive
3. Disease duration (since diagnosis) <10 years
4. Expanded Disability Status Scale (EDSS) at baseline 0-5.5
5. Untreated patients or patients being off therapy for the time-periods listed under exclusion criterion No. 2. Patients are either not eligible to receive approved therapies or have explicitly chosen not to receive such therapies after being adequately informed by the investigators
6. Only for female patients of childbearing potential (sexually mature, pre-menopausal and not surgically sterile): the patient is willing to use a highly effective method of contraception throughout the treatment phase or at least for 4 weeks after the last dose of the study drug
7. Male patients willing to use contraception (such as a condoms) throughout the treatment phase or at least for 4 weeks after the last dose of the study drug, unless surgically steril

Exclusion Criteria:

1. Patients with an active chronic disease (or stable but treated with immunomodulatory/-suppressive therapy) of the immune system other than MS (e.g. rheumatoid arthritis, scleroderma, Crohn's disease, ulcerative colitis, etc.) or with a known immunodeficiency syndrome (AIDS, hereditary immune deficiency, drug-induced immune deficiency)
2. Prior treatment with any of the medications specified in the protocol
3. History of HIV, chronic or active Hepatitis, chronic or active Hepatitis B or Syphilis
4. Long-Covid19 syndrome
5. History of splenectomy or chronic liver disease
6. History of coronary artery disease, chronic heart failure, aortic stenosis
7. Current anticoagulation therapy
8. Uncontrolled grade II hypertension (≥160 systolic and/or ≥100 diastolic blood pressure according to the International Society of Hypertension (ISH) guidelines) despite treatment or without treatment
9. History of stroke
10. Pregnant female confirmed by a positive pregnancy test or breast-feeding
11. History of alcohol or drug abuse within the 1 year prior to screening visit 1
12. History of or existing malignancy within the last 5 years prior to enrolment except history of basal cell carcinoma and melanoma in situ
13. History of or existing relevant central nervous system disorder (other than MS)
14. Allergy to gadolinium-based contrast agents
15. Any other disease or condition, which could interfere with the participation in the study according to the study protocol, or with the ability of the patients to cooperate and comply with the study procedures.
16. Anemia, defined as hemoglobin levels ≤12.5 g/dl (7.25 mmol/l) for female and ≤13.5 g/dl (8.37 mmol/l) for male participants (may be repeated if 11.5-12.5 g/dl in females and 12.5-13.5 g/dl in males)
17. Erythrocyte count <4.0 E12/L in female and <4.5 E12/L in male patients (may be repeated if >3.8 E12/L in female and >4.3 E12/L in male)
18. Lymphopenia with total lymphocyte counts ≤1000/µl (may be repeated if >800/µl)
19. Positive HIV testing
20. Positive results of baseline period testing for serological markers for hepatitis B, C, and Syphilis indicating acute or chronic infection
21. Patient is not eligible for blood donation according to local regulations
22. Having one or more of the following laboratory results:

    1. Estimated glomerular filtration rate (eGFR)< 60 mL/min/1.73 m2 (may be repeated if eGFR 45-59 mL/min/1.73 m2)
    2. ALT or AST >3x upper limit of normal (ULN; may be repeated if 3.1-4x ULN)
    3. Total bilirubin greater than 2x ULN (may be repeated if 2.1-3x ULN), with the exception for patients with Gilbert's disease
    4. Platelet count ≤100x109/L (may be repeated if 80-100x 109/L)
    5. Abnormalities in hepatic synthetic function tests as judged by the Investigator to be clinically significant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events as assessed by CTCAE v4.0 and worsening of MS [Safety of CLS12311] | on average 48 weeks
  Number and severity of adverse events (AEs) and serious adverse events (SAEs) and worsening of disease measured by clinical (relapses) and imaging (number & size of brain MRI lesions)

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events as assessed by CTCAE v4.0 in each dose group [Safety of CLS12311] | on average 48 weeks
  Number and severity of treatment-emergent AEs (TEAEs) and treatment-emergent SAEs (TESAEs) in each dose group
Incidence of patients experiencing worsening of MS in each dose group [Safety of CLS12311] | on average 48 weeks
  Number of confirmed relapses in the treatment phase in each dose group
Incidence of patients experiencing worsening of EDSS in each dose group [Safety of CLS12311] | on average 48 weeks
  Change in Expanded Disability Status Scale (EDSS) in each dose group
Incidence of patients experiencing worsening of T25-FW in each dose group [Safety of CLS12311] | on average 48 weeks
  Change in Timed 25-Foot Walk (T25-FW) in each dose group
Incidence of patients experiencing worsening of 9-HPT in each dose group [Safety of CLS12311] | on average 48 weeks
  Change in 9-Hole Peg Test (9-HPT) in each dose group
Incidence of patients experiencing worsening of SDMT in each dose group [Safety of CLS12311] | on average 48 weeks
  Change in Symbol Digit Modalities Test (SDMT) in each dose group

CONTACTS AND LOCATIONS:
Locations (8):
- Czechia (2):
  - RS Centrum - Neurologická klinika, Prague
  - Neurologická klinika 2. LF UK a FN Motol, Prague
- Germany (3):
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Klinik für Neurologie, Hamburg, Hamburg
  - Fraunhofer Institut für Translationale Medizin und Pharmakologie (ITMP), Göttingen, Lower Saxony
  - Universitätsklinikum Münster (UKM), Klinik für Neurologie, Münster, North Rhine-Westphalia
- Azienda Ospedaliero Universitaria Careggi, Florence, Tuscany, Italy
- Switzerland (2):
  - Bellevue Medical Group (BMG), Neurozentrum, Zurich, Canton of Zurich
  - UniversitätsSpital Zürich (USZ), Klinik für Neurologie, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: No